CLINICAL TRIAL: NCT05269407
Title: The Ability of the Change in Positional Perfusion Index in Predicting Post-spinal Anesthesia Hypotension in Caesarian Section
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mohamed abdelghany ali, Lecturer of anesthesia, Cairo University
Other Study IDs: N120
Record Dates: First submitted 2022-02-26; First posted 2022-03-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Obstetric Anesthesia Problems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Peripheral perfusion index — The study aimed to generate a model relating pre-spinal perfusion index to the likelihood and severity of the reduction in blood pressure in the first 20 min after spinal injection.
  A correlation between the delta PI and the delta SBP (the difference between the baseline maternal systolic blood pressure and the lowest blood pressure)will be investigated to establish a predictive model to define cut-off values at which perfusion index variation indicated a low risk (no or mild hypotension groups) or a high risk (moderate, severe groups) of reduction in blood pressure.. The incremental change of a measure PI, the ΔPI will be calculated as the absolute change in PI between supine and sitting positions, ΔPI=PIsupine-sitting. The relative change in PI the rPI, will be expressed as the percentage of change in PI, rPI=ΔPI/PIsitting× 100.

SUMMARY:
Our study aims to investigate the value of postural perfusion index changes as a non-invasive method to predict hypotension following spinal anesthesia for elective cesarean delivery.

DETAILED DESCRIPTION:
The perfusion index is the ratio of pulsatile blood flow to non-pulsatile in peripheral tissues and can be measured non-invasively using a pulse oximeter .Perfusion index measurement is considered a non-invasive rapid indicator of microcirculation variation and can help to detect circulation disturbance.It also can assess peripheral perfusion dynamics resulting from changes in peripheral vascular tone. Perfusion index changes according to posture with its highest value in Trendelenburg position and lowest value during 45-degree sitting position. However, to the best of our knowledge, no studies have studied the effect of posture on perfusion index in a full-term pregnancy, and its ability to predict hypotension following spinal anesthesia for elective cesarean delivery.

A previous study had found a correlation between baseline perfusion index and the incidence of post-spinal hypotension in the cesarean section, however, they haven't studied the effect of postural change on PI and its predictability of post-spinal induced hypotension(,Our study aims to investigate the value of postural perfusion index changes as a non-invasive method to predict hypotension following spinal anesthesia for elective cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1-2 Age > 18 years uncomplicated singleton pregnancy at full-term Elective scheduled caesarian section under spinal anesthesia

Exclusion Criteria:

* pre-existing hypertension gestational hypertension or preeclampsia Diabetes mellitus, or autonomic neuropathy Patients with peripheral vascular diseases known fetal abnormality. Emergency caesarian section. Placenta previa or placenta accrete. absolute contraindications or failure to perform spinal anesthesia.Study

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: A total of 115 consecutive adult female patients, aged >18 years scheduled for the elective caesarian section under spinal anesthesia will be included in the study.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2022-03-20 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Sensitivity of positional index in predicting post-spinal hypotension | 30 minutes post spinal anesthesia
  The sensitivity of perfusion index postural change in predicting post-spinal anesthesia hypotension in caesarian section. surgeries.

SECONDARY OUTCOMES:
The sensitivity of sitting perfusion index to predict post-spinal anesthesia hypotension in caesarian section. | 30 minutes post spinal anesthesia
  The sensitivity of sitting perfusion index to predict post-spinal anesthesia hypotension in caesarian section.
The sensitivity of supine perfusion index to predict post-spinal anesthesia hypotension in caesarian section. | 30 minutes post spinal anesthesia
  The sensitivity of sitting perfusion index to predict post-spinal anesthesia hypotension in caesarian section.
The correlation between perfusion index postural change and the degree of severity of hypotension in caesarian section post spina anesthesia. | 30 minutes post spinal anesthesia
  The correlation between perfusion index postural change and the degree of severity of hypotension in caesarian section post spina anesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided